CLINICAL TRIAL: NCT05188105
Title: Interventional Cross-over Study to Evaluate the Efficacy of Transcranial Alternating Current Stimulation (tACS) on Cognitive Performance in Patients With Dementia With Lewy Bodies
Brief Title: Alpha tACS in Dementia With Lewy Bodies
Acronym: Alpha-DLB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Responsible Party: Principal Investigator, Barbara Borroni, Clinical Professor, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NP4758
Record Dates: First submitted 2021-11-14; First posted 2022-01-12 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Dementia With Lewy Bodies; Lewy Body Disease
Keywords: Dementia with Lewy bodies; Lewy Body Disease; Alpha stimulation; transcranial alternating current stimulation
MeSH Terms: conditions — Lewy Body Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- real tACS (Experimental): Single session of alpha tACS (12 Hz) at 3 mA over the occipital cortex.
  Interventions: Device: Alpha tACS (12 Hz) over the occipital cortex
- sham tACS (Placebo Comparator): Single session of sham tACS over the occipital cortex.
  Interventions: Device: Alpha tACS (12 Hz) over the occipital cortex

INTERVENTIONS:
Device: Alpha tACS (12 Hz) over the occipital cortex — Single session of alpha tACS (12 Hz) over the occipital cortex

SUMMARY:
Brain oscillations are ubiquitous in the human brain and have been implicated in cognitive and behavioral states defined in precisely tuned neural networks. In neurodegenerative disorders, neurodegeneration is accompanied by changes in oscillatory activity leading to the emerging concept of neurological and psychiatric disorders as "oscillopathies".

Dementia with Lewy bodies (DLB), which is the second most frequent cause of neurodegenerative dementia, is characterized by an important alteration of brain oscillations. The restoration of oscillations by neuronal entrainment in animal models of neurodegenerative disease has shown a significant reduction in the neuropathological load of toxic proteins, with a consequent significant increase in cognitive performance.

Transcranial alternating current brain stimulation (tACS), is a neurophysiological method of non-invasive modulation of the excitability of the central nervous system that is having an increasingly numerous spectrum of potential therapeutic applications. Recent studies have demonstrated the effectiveness of this method in modulating the natural frequencies of cerebral oscillation, underlying multiple cognitive processes such as verbal memory, perception and working memory.

On the basis of these premises, the treatment with alpha tACS is proposed in patients with DLB.

In this randomized, double-blind, sham-controlled, cross-over study, the investigators will evaluate whether a single stimulation with alpha tACS on the occipital lobes can improve symptoms in patients with DLB.

DETAILED DESCRIPTION:
Brain oscillations are ubiquitous in the human brain and have been implicated in cognitive and behavioral states defined in precisely tuned neural networks. In neurodegenerative disorders, neurodegeneration is accompanied by changes in oscillatory activity leading to the emerging concept of neurological and psychiatric disorders as "oscillopathies".

Dementia with Lewy bodies (DLB), which is the second most frequent cause of neurodegenerative dementia, is characterized by an important alteration of brain oscillations. The restoration of oscillations by neuronal entrainment in animal models of neurodegenerative disease has shown a significant reduction in the neuropathological load of toxic proteins, with a consequent significant increase in cognitive performance.

Transcranial alternating current brain stimulation (tACS), is a neurophysiological method of non-invasive modulation of the excitability of the central nervous system that is having an increasingly numerous spectrum of potential therapeutic applications. Recent studies have demonstrated the effectiveness of this method in modulating the natural frequencies of cerebral oscillation, underlying multiple cognitive processes such as verbal memory, perception and working memory.

On the basis of these premises, the treatment with alpha tACS is proposed in patients with DLB.

In this randomized, double-blind, sham-controlled, cross-over study, the investigators will evaluate whether a single stimulation with alpha tACS on the occipital lobes can improve symptoms in patients with DLB.

Subjects will be randomized in two groups, one receiving a single treatment with alpha tACS (12 Hz) first and the other receiving sham stimulation. After one week the treatments will be exchanged. Patients will be evaluated with neuropsychological tests and neurophysiological measures of cholinergic transmission.

ELIGIBILITY:
Inclusion Criteria:

* Dementia with Lewy bodies (criteria according to McKeith, Neurology 2017).

Exclusion Criteria:

* Cerebrovascular disorders, previous stroke, hydrocephalus, and intra-cranial mass documented by MRI.
* History of traumatic brain injury or other neurological diseases.
* Serious medical illness other than DLB
* History of seizures
* Pregnancy
* Metal implants in the head (except dental fillings)
* Electronic implants (i.e. pace-maker, implanted medical pump)
* Age <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2024-03-10 (Actual); Study Completion 2024-03-20 (Actual)

PRIMARY OUTCOMES:
Changes in Visual Search Task Test scores | 40 minutes after the start of the intervention
  The visual search task requires participants to determine whether a target (such as a particular letter, shape, or image) is present in an array of other stimuli. The task consists of two parts, each with 64 stimuli, for a total of 128 stimuli. Participants are asked to look at the screen and press a button if the target stimulus is present or another button if the target stimulus is absent. After pressing the chosen button, a feedback will appear on the screen that will tell the subject if his answer is correct or incorrect. Subjects must respond as quickly as possible, otherwise the answer will be considered missed and they will proceed to the next screen.
  The score ranges from 0 (worse performance) to 128 (best performance).

SECONDARY OUTCOMES:
Changes in Rey Auditory Verbal Learning Test scores | Baseline (immediately before the intervention) - Immediately after the intervention
  Participants are given a list of 15 unrelated words repeated over five different trials and are asked to repeat. Another list of 15 unrelated words are given and the patient must again repeat the original list of 15 words and then again after 30 minutes.
  The score ranges from 0 (worse performance) to 15 (best performance).
Changes in Trail Making Test Part A | Baseline (immediately before the intervention) - Immediately after the intervention
  The Trail Making Test Part A consists of 25 circles on a piece of paper with the numbers 1-25 written randomly in the circles. The test taker's task is to start with number one and draw a line from that circle to the circle with the number two in it to the circle with the three in it, etc. The person continues to connect the circles in numerical order until they reach number 25.
  Scoring is based on time taken to complete the test with lower scores being better.
Changes in Trail Making Test Part B | Baseline (immediately before the intervention) - Immediately after the intervention
  The Trail Making Test Part B consists of 24 circles on a piece of paper, but rather than all of the circles containing numbers, half of the circles have the numbers 1-12 in them and the other half (12) contain the letters A-L. The person taking the test has to draw a line from one circle to the next in ascending order; however, he must alternate the circles with numbers in them (1-13) with circles with letters in them (A-L). In other words, he is to connect the circles in order like this: 1-A-2-B-3-C-4-D-5-E and so on.
  Scoring is based on time taken to complete the test with lower scores being better.
Changes in relative alpha power in occipital EEG leads | Baseline (immediately before the intervention) - Immediately after the intervention
  By using electroencephalography (EEG), the investigators will evaluate the effects of alpha tACS on relative alpha power in occipital EEG leads.
Change in SAI measurements | Baseline (immediately before the intervention) - Immediately after the intervention
  By using transcranial magnetic stimulation (TMS), the investigators will evaluate the effects of alpha tACS on short latency afferent inhibition (SAI), which is a marker of cholinergic transmission.
Change in SICI measurements | Baseline (immediately before the intervention) - Immediately after the intervention
  By using transcranial magnetic stimulation (TMS), the investigators will evaluate the effects of alpha tACS on short interval intracortical inhibition (SICI), which is a marker of GABAergic transmission.
Change in ICF measurements | Baseline (immediately before the intervention) - Immediately after the intervention
  By using transcranial magnetic stimulation (TMS), the investigators will evaluate the effects of alpha tACS on intracortical facilitation (ICF), which is a marker of glutamatergic transmission.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Borroni, MD, Principal Investigator — ASST Spedali Civili di Brescia; Alberto Benussi, MD, Principal Investigator — ASST Spedali Civili di Brescia
Locations (1):
- ASST Spedali Civili di Brescia, Brescia, BS, Italy

IPD SHARING:
Plan to Share IPD: Yes
All data, including outcome measure results, study protocol and statistical analysis plan, will be shared upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the study completion indefinitely.
Access Criteria: Reasonable request

REFERENCES:
- [Background] McKeith IG, Boeve BF, Dickson DW, Halliday G, Taylor JP, Weintraub D, Aarsland D, Galvin J, Attems J, Ballard CG, Bayston A, Beach TG, Blanc F, Bohnen N, Bonanni L, Bras J, Brundin P, Burn D, Chen-Plotkin A, Duda JE, El-Agnaf O, Feldman H, Ferman TJ, Ffytche D, Fujishiro H, Galasko D, Goldman JG, Gomperts SN, Graff-Radford NR, Honig LS, Iranzo A, Kantarci K, Kaufer D, Kukull W, Lee VMY, Leverenz JB, Lewis S, Lippa C, Lunde A, Masellis M, Masliah E, McLean P, Mollenhauer B, Montine TJ, Moreno E, Mori E, Murray M, O'Brien JT, Orimo S, Postuma RB, Ramaswamy S, Ross OA, Salmon DP, Singleton A, Taylor A, Thomas A, Tiraboschi P, Toledo JB, Trojanowski JQ, Tsuang D, Walker Z, Yamada M, Kosaka K. Diagnosis and management of dementia with Lewy bodies: Fourth consensus report of the DLB Consortium. Neurology. 2017 Jul 4;89(1):88-100. doi: 10.1212/WNL.0000000000004058. Epub 2017 Jun 7. PMID 28592453
- [Background] Franciotti R, Pilotto A, Moretti DV, Falasca NW, Arnaldi D, Taylor JP, Nobili F, Kramberger M, Ptacek SG, Padovani A, Aarlsand D, Onofrj M, Bonanni L; E-DLB consortium. Anterior EEG slowing in dementia with Lewy bodies: a multicenter European cohort study. Neurobiol Aging. 2020 Sep;93:55-60. doi: 10.1016/j.neurobiolaging.2020.04.023. Epub 2020 Apr 29. PMID 32450445
- [Background] Aoki Y, Kazui H, Pascal-Marqui RD, Ishii R, Yoshiyama K, Kanemoto H, Suzuki Y, Sato S, Hata M, Canuet L, Iwase M, Ikeda M. EEG Resting-State Networks in Dementia with Lewy Bodies Associated with Clinical Symptoms. Neuropsychobiology. 2019;77(4):206-218. doi: 10.1159/000495620. Epub 2019 Jan 17. PMID 30654367
- [Background] Schumacher J, Thomas AJ, Peraza LR, Firbank M, Cromarty R, Hamilton CA, Donaghy PC, O'Brien JT, Taylor JP. EEG alpha reactivity and cholinergic system integrity in Lewy body dementia and Alzheimer's disease. Alzheimers Res Ther. 2020 Apr 22;12(1):46. doi: 10.1186/s13195-020-00613-6. PMID 32321573
- [Background] Schumacher J, Taylor JP, Hamilton CA, Firbank M, Cromarty RA, Donaghy PC, Roberts G, Allan L, Lloyd J, Durcan R, Barnett N, O'Brien JT, Thomas AJ. Quantitative EEG as a biomarker in mild cognitive impairment with Lewy bodies. Alzheimers Res Ther. 2020 Jul 8;12(1):82. doi: 10.1186/s13195-020-00650-1. PMID 32641111
- [Background] Bonanni L, Franciotti R, Nobili F, Kramberger MG, Taylor JP, Garcia-Ptacek S, Falasca NW, Fama F, Cromarty R, Onofrj M, Aarsland D; E-DLB study group. EEG Markers of Dementia with Lewy Bodies: A Multicenter Cohort Study. J Alzheimers Dis. 2016 Oct 18;54(4):1649-1657. doi: 10.3233/JAD-160435. PMID 27589528
- [Background] Pascarelli MT, Del Percio C, De Pandis MF, Ferri R, Lizio R, Noce G, Lopez S, Rizzo M, Soricelli A, Nobili F, Arnaldi D, Fama F, Orzi F, Buttinelli C, Giubilei F, Salvetti M, Cipollini V, Franciotti R, Onofri M, Fuhr P, Gschwandtner U, Ransmayr G, Aarsland D, Parnetti L, Farotti L, Marizzoni M, D'Antonio F, De Lena C, Guntekin B, Hanoglu L, Yener G, Emek-Savas DD, Triggiani AI, Paul Taylor J, McKeith I, Stocchi F, Vacca L, Hampel H, Frisoni GB, Bonanni L, Babiloni C. Abnormalities of resting-state EEG in patients with prodromal and overt dementia with Lewy bodies: Relation to clinical symptoms. Clin Neurophysiol. 2020 Nov;131(11):2716-2731. doi: 10.1016/j.clinph.2020.09.004. Epub 2020 Sep 23. PMID 33039748
- [Background] van Dellen E, de Waal H, van der Flier WM, Lemstra AW, Slooter AJ, Smits LL, van Straaten EC, Stam CJ, Scheltens P. Loss of EEG Network Efficiency Is Related to Cognitive Impairment in Dementia With Lewy Bodies. Mov Disord. 2015 Nov;30(13):1785-93. doi: 10.1002/mds.26309. Epub 2015 Jul 16. PMID 26179663
- [Background] Briel RC, McKeith IG, Barker WA, Hewitt Y, Perry RH, Ince PG, Fairbairn AF. EEG findings in dementia with Lewy bodies and Alzheimer's disease. J Neurol Neurosurg Psychiatry. 1999 Mar;66(3):401-3. doi: 10.1136/jnnp.66.3.401. PMID 10084544
- [Background] Bonanni L, Thomas A, Tiraboschi P, Perfetti B, Varanese S, Onofrj M. EEG comparisons in early Alzheimer's disease, dementia with Lewy bodies and Parkinson's disease with dementia patients with a 2-year follow-up. Brain. 2008 Mar;131(Pt 3):690-705. doi: 10.1093/brain/awm322. Epub 2008 Jan 17. PMID 18202105
- [Background] Massa F, Meli R, Grazzini M, Fama F, De Carli F, Filippi L, Arnaldi D, Pardini M, Morbelli S, Nobili F. Utility of quantitative EEG in early Lewy body disease. Parkinsonism Relat Disord. 2020 Jun;75:70-75. doi: 10.1016/j.parkreldis.2020.05.007. Epub 2020 May 24. PMID 32480310
- [Background] Dauwan M, van Dellen E, van Boxtel L, van Straaten ECW, de Waal H, Lemstra AW, Gouw AA, van der Flier WM, Scheltens P, Sommer IE, Stam CJ. EEG-directed connectivity from posterior brain regions is decreased in dementia with Lewy bodies: a comparison with Alzheimer's disease and controls. Neurobiol Aging. 2016 May;41:122-129. doi: 10.1016/j.neurobiolaging.2016.02.017. Epub 2016 Feb 21. PMID 27103525
- [Background] Babiloni C, Del Percio C, Lizio R, Noce G, Lopez S, Soricelli A, Ferri R, Nobili F, Arnaldi D, Fama F, Aarsland D, Orzi F, Buttinelli C, Giubilei F, Onofrj M, Stocchi F, Stirpe P, Fuhr P, Gschwandtner U, Ransmayr G, Garn H, Fraioli L, Pievani M, Frisoni GB, D'Antonio F, De Lena C, Guntekin B, Hanoglu L, Basar E, Yener G, Emek-Savas DD, Triggiani AI, Franciotti R, Taylor JP, Vacca L, De Pandis MF, Bonanni L. Abnormalities of resting-state functional cortical connectivity in patients with dementia due to Alzheimer's and Lewy body diseases: an EEG study. Neurobiol Aging. 2018 May;65:18-40. doi: 10.1016/j.neurobiolaging.2017.12.023. Epub 2017 Dec 30. PMID 29407464
- [Background] Babiloni C, Del Percio C, Lizio R, Noce G, Cordone S, Lopez S, Soricelli A, Ferri R, Pascarelli MT, Nobili F, Arnaldi D, Aarsland D, Orzi F, Buttinelli C, Giubilei F, Onofrj M, Stocchi F, Stirpe P, Fuhr P, Gschwandtner U, Ransmayr G, Caravias G, Garn H, Sorpresi F, Pievani M, Frisoni GB, D'Antonio F, De Lena C, Guntekin B, Hanoglu L, Basar E, Yener G, Emek-Savas DD, Triggiani AI, Franciotti R, De Pandis MF, Bonanni L. Abnormalities of cortical neural synchronization mechanisms in patients with dementia due to Alzheimer's and Lewy body diseases: an EEG study. Neurobiol Aging. 2017 Jul;55:143-158. doi: 10.1016/j.neurobiolaging.2017.03.030. Epub 2017 Apr 5. PMID 28454845
- [Background] Tavakoli AV, Yun K. Transcranial Alternating Current Stimulation (tACS) Mechanisms and Protocols. Front Cell Neurosci. 2017 Sep 1;11:214. doi: 10.3389/fncel.2017.00214. eCollection 2017. PMID 28928634
- [Background] Klink K, Passmann S, Kasten FH, Peter J. The Modulation of Cognitive Performance with Transcranial Alternating Current Stimulation: A Systematic Review of Frequency-Specific Effects. Brain Sci. 2020 Dec 2;10(12):932. doi: 10.3390/brainsci10120932. PMID 33276533